CLINICAL TRIAL: NCT00599820
Title: OCT, Visual Outcome and Angiographic Analysis of Choroidal Neovascularization in Six Eyes With Angioid Streaks Treated With a Single Intravitreal Injection of Bevacizumab
Brief Title: Use of Intravitreal Bevacizumab in Eyes With Choroidal Neovascularization Secondary to Angioid Streaks
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC 010
Record Dates: First submitted 2006-06-30; First posted 2008-01-24 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Angioid Streaks; Choroidal Neovascularization
Keywords: Angioid Streaks; Choroidal Neovascularization; Bevacizumab
MeSH Terms: conditions — Angioid Streaks; Choroidal Neovascularization

INTERVENTIONS:
Drug: Intravitreal Bevacizumab

SUMMARY:
Intravitreal Bevacizumab is an effective treatment for choroidal neovascularization secondary to Angioid Streaks

DETAILED DESCRIPTION:
A consecutive case series of patients with angioid streaks that developed subfoveal choroidal neovascularization were treated with a primary 2.5 mg injection of Bevacizumab (Avastin) intravitreally. All patients were evaluated with BCVA at 1, 2 , 4 and 12 weeks and OCT and fluoresceine angiography at month 1 and 3. (Patients will be follow 6 months)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Angioid Streaks
* Choroidal neovascularization associated
* Untreated patients or patients treated once with PDT

Exclusion Criteria:

* Ocular surgery excepting uncomplicated phacoemulsification
* Glaucoma or any other ocular pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-11 (Actual); Primary Completion 2005-11 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
BCVA
Fluoresceine Angiography
Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Solís-Vivanco, MD, Principal Investigator — Asociación para Evitar la Ceguera en México; Jans Fromow-Guerra, MD PhD, Study Chair — Asociación para Evitar la Ceguera en México; Mariana Martínez-Castellanos, MD, Study Chair — Asociación para Evitar la Ceguera en México; Elizabeth Reyna-Castelán, MD, Study Chair — Asociación para Evitar la Ceguera en México; Myriam Hernández-Rojas, MD, Study Chair — Asociación para Evitar la Ceguera en México; Griselda Alvarez-Rivera, MD, Study Chair — Asociación para Evitar la Ceguera en México; Hugo Quiroz-Mercado, MD, Study Director — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México (APEC), Mexico City, Mexico City, Mexico